CLINICAL TRIAL: NCT01379638
Title: Best Cardiac Output During Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Sisse Anette Thomassen, Department of cardiothoracic surgery and anesthesiology
Other Study IDs: N-20080035
Record Dates: First submitted 2011-06-22; First posted 2011-06-23 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2008-12

CONDITIONS: Bypass Complications
Keywords: cardiopulmonary bypass; cardiac output; flow rate; lactate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cardiac output: Adult patients undergoing cardiac surgery with normothermic cardiopulmonary bypass

SUMMARY:
The purpose of this study is to determine whether the patients cardiac output measured before cardiopulmonary bypass (CPB), is more sufficient to secure the patients oxygen needs than the estimated cardiac output from Ficks principle, and thereby prevent organ failure.

DETAILED DESCRIPTION:
For more than 50 years, CPB has been used to mechanically support the functions of the heart and lungs. In early studies, systemic oxygen uptake, calculated using Ficks global principle, was used to assess the efficiency of CPB. Using this measure of efficiency, a pump flow rate in liters per minute, based on the product of the body surface area (BSA) and a constant of 2.4 was found adequate to perfuse the body during normothermia. Ficks global principle is still used together with other methods to secure adequated perfusion under CPB.

The purpose of this study is to determine whether the patients cardiac output measured before CPB, is more sufficient to secure the patients oxygen needs than the estimated cardiac output from Ficks principle, and thereby prevent organ failure.

The hypothesis is that the patients cardiac output is a better marker for the optimal cardiac output than the estimated cardiac output.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted for scheduled cardiac surgery during cardiopulmonary bypass
* Aged 18-90 years
* LVEF > 50 %
* written consent from the patients

Exclusion Criteria:

* Former cerebral emboli
* Former head trauma
* known stenosis of the arteria carotis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients to be admitted to Aalborg Hospital, department of cardiac surgery for scheduled cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bodil Steen Rasmussen, MD, PhD, Study Director — Aalborg University Hospital
Locations (1):
- Alborg Hospital, Aalborg, Aalborg, Denmark